CLINICAL TRIAL: NCT03132792
Title: A Phase I Open Label Clinical Trial Evaluating the Safety and Anti-Tumor Activity of Autologous T Cells Expressing Enhanced TCRs Specific for Alpha Fetoprotein (AFPᶜ³³²T) in HLA-A2 Positive Subjects With Advanced Hepatocellular Carcinoma (HCC) or Other AFP Expressing Tumor Types
Brief Title: AFPᶜ³³²T in Advanced HCC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Adaptimmune (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADP-0033-001; 2017-000778-12 (EudraCT Number)
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Cancer; AFP Expressing Tumors
Keywords: Alpha-fetoprotein; Cell Therapy; T Cell Therapy; SPEAR T Cell; Immuno-oncology; Metastatic; Previously treated; T Cell Receptor
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous genetically modified AFPᶜ³³²T cells (Experimental)
  Interventions: Genetic: Autologous genetically modified AFPᶜ³³²T cells

INTERVENTIONS:
Genetic: Autologous genetically modified AFPᶜ³³²T cells — Infusion of autologous genetically modified AFPᶜ³³²T cells

SUMMARY:
This first time in human study is intended for men and women between 18 and 75 years of age who have advanced liver cancer which has grown or returned after being treated or another AFP expressing tumor. Those who did not tolerate or refused other therapies may also participate. The purpose of this study is to test the safety of genetically changed T cells that target alpha-fetoprotein (AFP) and find out what effects, if any, they have in subjects with liver cancer or other AFP expressing tumor types. This study is for subjects who have a blood test positive for appropriate HLA-A*02 P Group and have adequate AFP protein in blood or tumor, and whose noncancerous liver tissue has very little AFP protein (Liver only).

The study will take the subject's T cells, which are a natural type of immune cell in the blood, and send them to a laboratory to be modified. The changed T cells used in this study will be the subject's own T cells that have been genetically changed with the aim of attacking and destroying cancer cells.

The manufacturing of T cells takes about 1 month to complete. The T cells will be given back to the subject through an intravenous infusion after 3 days of chemotherapy. The study will evaluate three different cell dose levels in order to find out the target cell dose. Once the target cell dose is determined, additional subjects will be enrolled to further test the safety and effects at this cell dose.

Subjects will be hospitalized for at least 1 week after receiving their T cells back and then seen frequently by the Study Physician for the next 6 months. After that, subjects will be seen every three months. If subjects have disease progression or withdraw from the study, they will then be entered into a long-term follow up for safety monitoring. In long-term follow up, subjects will be seen every 6 months by their Study Physician for the first 5 years after the T cell infusion and annually for the next 10 years.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject is ≥ 18 years and ≤ 75 years of age and has voluntarily agreed to participate by giving written informed consent in accordance with ICH GCP Guidelines and applicable local regulations.
2. Histologically confirmed HCC, not amenable to transplant, resection. Subjects may undergo loco-regional therapy after enrollment but not at time of lymphodepletion. Or Histologically confirmed diagnosis of another AFP expressing tumor (e.g. cholangiocarcinoma).
3. Measurable disease according to RECIST 1.1 criteria prior to lymphodepletion.
4. Progressive disease following or intolerant of or refuses standard of care systemic therapy prior to lymphodepletion.
5. Positive for any A*02:01 P group allele.
6. a) Group 1, 2, 3, (HCC) Subjects will be eligible for enrollment if they meet either one of these AFP expression criteria:

   * AFP expression of ≥1+ in ≥20% of tumor cells by immunohistochemistry and their non-cancerous liver tissue has ≤5% cells stained for AFP at any intensity by immunohistochemistry.
   * Serum AFP levels of ≥100ng/mL and their non-cancerous liver tissue has ≤5% cells stained for AFP at any intensity by immunohistochemistry.

6. b) Group 4 (other AFP expressing tumor types) Subjects will be eligible for enrollment if they meet either one of these AFP expression criteria:

o Serum AFP levels of ≥100ng/mL and their non-cancerous liver tissue (if applicable) has ≤5% cells stained for AFP at any intensity by immunohistochemistry.

7. Life expectancy of > 4 months 8. Child-Pugh score ≤ 6 9. Eastern Cooperative Oncology Group (ECOG) 0-1 10. Subject must have adequate organ function as defined in the protocol.

Key Exclusion Criteria:

1. Positive for any of the HLA-A*02 allele other than HLA-A*02:01 P Group, HLA-A*02:03 P group or null alleles or positive for the following alleles: HLA-C*04:04 or HLA-B*51:03.
2. Prior liver transplant
3. Received the following prior to leukapheresis:

   1. Cytotoxic chemotherapy, immune therapy and biological therapy within 3 weeks
   2. Corticosteroids or any other immunosuppressive therapy within 2 weeks. NOTE: Use of inhaled or topical steroids is not exclusionary
   3. Sorafenib/Regorafenib/Lenvatinib within 1 week
   4. Cabozantinib within 2 weeks
   5. Duration of treatment free intervals for any other anti-cancer therapies must be discussed with Adaptimmune Study Physician.
4. Received the following prior to lymphodepleting chemotherapy :

   1. Cytotoxic chemotherapy or loco-regional therapy within 3 weeks, liver directed radiation therapy within three months.
   2. Corticosteroids or any other immunosuppressive therapy within 2 weeks. NOTE: Use of inhaled or topical steroids is not exclusionary
   3. Bone/soft tissue directed palliative radiotherapy within 4 weeks.
   4. Investigational treatment or clinical trial within 4 weeks.
   5. Sorafenib/Regorafenib/Lenvatinib within 1 week.
   6. Cabozantinib within 2 weeks
   7. Prior cancer-directed immunotherapy within 4 weeks, including monoclonal antibodies against PD-1 receptor or ligand.
   8. Use of an experimental vaccine within 2 months in the absence of tumor response. The subject should be excluded if their disease is responding to an experimental vaccine given within 6 months
   9. Any previous gene therapy using an integrated vector
   10. Duration of treatment free intervals for any other anti-cancer therapies must be discussed with Adaptimmune Study Physician.
5. Toxicity persisting from previous anti-cancer therapy of ≥ Grade 2 (except for non-clinically significant toxicities, e.g., alopecia, vitiligo). Subjects with Grade 2 toxicities that are deemed stable or irreversible (e.g. peripheral neuropathy) can be enrolled on a case-by-case basis with prior consultation and agreement with the Sponsor Study Physician.
6. Major surgery within 4 weeks prior to lymphodepletion; subjects should have been fully recovered from any surgical related toxicities.
7. Bleeding ≥ Grade 2 in the past 3 months prior to lymphodepletion
8. Therapeutic anticoagulation from lymphodepletion until platelet count recovery (prophylactic heparin allowed)
9. Clinically or radiographically detectable ascites (beyond trace/rim of ascites) or ascites requiring medication
10. Clinically detectable hepatic encephalopathy or hepatic encephalopathy requiring medication
11. Active viral hepatitis Subjects positive for hepatitis B surface antigen not on antiviral treatment/prophylaxis or subjects with detectable hepatitis B DNA

    1. Subjects with resolved (surface antigen negative, core antibody positive) or chronic stable (surface antigen positive) hepatitis B on antiviral treatment/prophylaxis with DNA levels of ≤100 IU/mL are allowed with HBV DNA monitoring after treatment
    2. Subjects with hepatitis C allowed provided they meet all other eligibility criteria
12. Positive serology for HIV
13. Positive serology for HTLV 1 or 2
14. History of chronic or recurrent (within the last year) severe autoimmune or immune mediated disease requiring steroids or other immunosuppressive treatments. Subjects with history of idiopathic autoimmune hepatitis are excluded. Subjects who experienced hepatitis during treatment with check point inhibiting antibodies are not excluded.
15. Subject has brain metastases.
16. Other active malignancy besides HCC or other eligible AFP expressing tumor types within 3 years.
17. Electrocardiogram (ECG) showing clinically significant abnormality at Screening or showing a QTc interval ≥450 msec in males and ≥470 msec in females (≥480 msec for subjects with Bundle Branch Block (BBB) over consecutive ECGs).
18. Bacterial or opportunistic infection within 3 months of treatment (upper respiratory infection and uncomplicated urinary tract infection allowed)
19. Uncontrolled intercurrent illness considered by the Investigator to add appreciable risk to study participation, including but not limited to:

    1. Clinically significant cardiac disease defined by CHF New York Heart Association (NYHA) > Class 1; uncontrolled clinically significant arrhythmia in last 6 months; Acute Coronary Syndrome (ACS) (angina or myocardial infarction) in last 6 months.
    2. Oxygen dependent lung disease.
    3. Clinically significant psychiatric illness/social situations that would limit compliance with study requirements.
    4. History of stroke or central nervous system bleeding; transient ischemic attack (TIA) or reversible ischemic neurologic deficit (RIND) in last 6 months.
20. Pregnant or breastfeeding
21. Alcohol or illicit drug dependency
22. Known contraindication to cyclophosphamide, fludarabine, mesna, G-CSF or other agents associated with study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2025-12-07 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with dose-limiting toxicity (DLT) and adverse events (AEs) and determination of optimally tolerated dose range, including serious adverse events (SAE). | 2 years
  Determine if treatment with autologous genetically modified T cells, (AFPᶜ³³²T) is safe and tolerable through assessment of DLTs, AEs, including SAEs; laboratory assessments including chemistry, hematology, coagulation, cardiac assessments including ECG, and cardiac Troponin

SECONDARY OUTCOMES:
Proportion of subjects with a confirmed Complete Response (CR) or Partial Response (PR) | 2 years
  Evaluation of the efficacy of the treatment by assessment of the Overall Response Rate according to RECIST v1.1
Interval between the date of first T cell infusion dose and first documented evidence of CR or PR | 2 years
  Evaluation of the efficacy of the treatment by assessment of time to first response
Interval between the date of first documented evidence of CR or PR until first documented disease progression or death due to any cause | 2 years
  Evaluation of the efficacy of the treatment by assessment of duration of response
Interval between the date of first documented evidence of SD until first documented disease progression or death due to any cause | 2 years
  Evaluation of the efficacy of the treatment by assessment of duration of stable disease
Interval between the date of first T cell infusion and the earliest date of disease progression or death due to any cause | 2 years
  Evaluation of the efficacy of the treatment by assessment of progression-free survival
Interval between the date of first T cell infusion and date of disease progression or death due to any cause | 2 years
  Evaluation of the efficacy of the treatment by assessment of overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Finn, MD, Principal Investigator — University of California, Los Angeles
Locations (21):
- United States (12):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - University of Miami, Miami, Florida
  - Winship Cancer Institute - Emory University, Atlanta, Georgia
  - University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic Clinical Trial Referral Office, Rochester, Minnesota
  - Washington University - School of Medicine, St Louis, Missouri
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Centre, Seattle, Washington
  - SCCA Immunotherapy Trials Intake, Seattle, Washington
- France (3):
  - Paoli Calmettes Institute, Marseille
  - Centre Eugène Marquis, Rennes
  - Institute Gustave Roussy, Villejuif
- Spain (2):
  - University Hospital of Barcelona, Barcelona
  - University Hospital of Navarra, Pamplona
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Guy's Hospital, London
  - NIHR UCLH Clinical Research, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meyer T, Finn RS, Borad M, Mahipal A, Edeline J, Houot R, Hausner PF, Hollebecque A, Goyal L, Frigault M, Evans TRJ, Wong KM, Tan BR, Mitry E, Sarker D, Feun L, El-Rayes B, Thistlethwaite F, Kaseb A, Alese O, Jin Z, Cirillo C, Bruix J, Roddie C, Noto P, Fayngerts S, Cristiani S, Sampson J, Bai J, Isabelle M, Broad R, Sun A, Norry E, Sangro B. Phase I trial of ADP-A2AFP TCR T-cell therapy in patients with advanced hepatocellular or gastric hepatoid carcinoma. J Hepatol. 2026 Jan;84(1):113-121. doi: 10.1016/j.jhep.2025.07.033. Epub 2025 Aug 12. PMID 40812667